CLINICAL TRIAL: NCT05904002
Title: Effect of Incentive Spirometery on Asthmatic Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Amin Soliman, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Eman_Amin_2023
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Asthmatic; Pregnant With Complication
MeSH Terms: conditions — Asthma; Pregnancy Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulmicort inhaler (Experimental): Group (A) consists of 30 patients. They will receive their inhaled glucocorticoids (pulmicort inhaler) on needs.
  Interventions: Drug: pulmicort inhaler
- incentive spirometer (Experimental): Group (B) consists of 30 patients. They will receive the same medical treatment and incentive spirometer program 3 days per week for six weeks.
  Interventions: Drug: pulmicort inhaler; Device: Incentive spirometer treatment

INTERVENTIONS:
Drug: pulmicort inhaler — Each woman in both groups (A&B) will receive pulmicort inhaler on needs.
Device: Incentive spirometer treatment — Each patient in group B will be instructed about the effects of incentive spirometer to gain their cooperation during the study course.
  Arms: incentive spirometer

SUMMARY:
The purpose of this study is to determine the effect of the incentive spirometer on asthma during pregnancy.

DETAILED DESCRIPTION:
This study will provide an evidence basis for obstetricians and physical therapist for women's health about the effect of spirometry on asthma during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

The patients will have the following criteria:

1. Their age will range from 30 to40years old.
2. Body mass index (BMI) will range from 25-29.9 kg/m2.
3. All patients will be clinically and medically stable.

Exclusion Criteria:

Patients will be excluded from the study if they have the following:

1. Diabetes mellitus.
2. Severe hypertension.
3. Neurological and neuromuscular disorders.
4. Blindness.
5. Developed moderate and severe degree of pleural effusion.
6. Cardiovascular instability.
7. Chronic chest disease.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Assessing the change in lung functions | at baseline and after 6 weeks of intervention
  The spirometer will be used for assessment of lung functions including total lung capacity (TLC) (litre), which is the most widely used functional index in the asthma follow up.
Assessing the change in symptoms of asthma | at baseline and after 6 weeks of intervention
  The Asthma Control Test provides a numerical score to help you and your healthcare provider determine if your asthma symptoms are well controlled. Take this test if you are 12 years or older. Share the score with your healthcare provider.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided